CLINICAL TRIAL: NCT00446199
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Determine the Lowest Effective Dose of Combinations of Oral Drospirenone and 17 Beta-Estradiol for the Relief of Moderate to Severe Vasomotor Symptoms in Postmenopausal Women Over a Treatment Period of 12 Weeks
Brief Title: Low-dose Hormone Therapy for Relief of Vasomotor Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91493; 310184 (Other: Company internal)
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Results first posted 2012-04-18 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Vasomotor Symptoms; Hot Flashes
Keywords: Vasomotor symptom relief; Postmenopausal women; Severe to Moderate Vasomotor symptoms
MeSH Terms: conditions — Hot Flashes | interventions — drospirenone; Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.5mg DRSP / 0.5mg E2 (BAY86-4891) (Experimental): One tablet [0.5mg drospirenone/0.5mg 17β-estradiol (DRSP/E2)] per day taken orally for 3 cycles (28 days per cycle).
  Interventions: Drug: 0.5mg DRSP / 0.5mg E2 (BAY86-4891)
- 0.25mg DRSP / 0.5mg E2 (BAY86-4891) (Experimental): One tablet [0.25mg drospirenone/0.5mg 17β-estradiol (DRSP/E2)] per day taken orally for 3 cycles (28 days per cycle).
  Interventions: Drug: 0.25mg DRSP / 0.5mg E2 (BAY86-4891)
- Estradiol (E2 0.3mg) (Experimental): One tablet [17β-estradiol (E2 0.3mg)] per day taken orally for 3 cycles (28 days per cycle).
  Interventions: Drug: Estradiol (E2 0.3mg)
- Placebo (Placebo Comparator): Matching placebo tablet per day taken orally for 3 cycles (28 days per cycle).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) — One tablet [0.5mg drospirenone/0.5mg 17β-estradiol (DRSP/E2)] per day taken orally for 3 cycles (28 days per cycle).
  Arms: 0.5mg DRSP / 0.5mg E2 (BAY86-4891)
Drug: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) — One tablet [0.25mg drospirenone/0.5mg 17β-estradiol (DRSP/E2)] per day taken orally for 3 cycles (28 days per cycle).
  Arms: 0.25mg DRSP / 0.5mg E2 (BAY86-4891)
Drug: Estradiol (E2 0.3mg) — One tablet [17β-estradiol (E2 0.3mg)] per day taken orally for 3 cycles (28 days per cycle).
  Arms: Estradiol (E2 0.3mg)
Drug: Placebo — Matching placebo tablet per day taken orally for 3 cycles (28 days per cycle).
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the lowest effective dose of the study drug for the relief of moderate to severe vasomotor symptoms in postmenopausal women for 12 weeks.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.

Bayer HealthCare Pharmaceuticals, Inc. is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

- Postmenopausal women >40 years of age experiencing a minimum of 7 to 8 moderate to severe hot flushes per day or 50 to 60 moderate to severe hot flushes per week

Exclusion Criteria:

* The usual exclusion criteria for hormone therapy apply
* Intake of medications other than hormones affecting hot flushes

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 735 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (67):
- United States (67):
  - Mobile, Alabama
  - Chandler, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Paramount, California
  - San Diego, California
  - Valley Village, California
  - Vista, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - New Britain, Connecticut
  - Boynton Beach, Florida
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Lake Worth, Florida
  - Leesburg, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Arlington Heights, Illinois
  - Champaign, Illinois
  - La Grange Park, Illinois
  - Newburgh, Indiana
  - Lexington, Kentucky
  - Amite, Louisiana
  - Marrero, Louisiana
  - Paw Paw, Michigan
  - Chaska, Minnesota
  - Springfield, Missouri
  - Billings, Montana
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Reno, Nevada
  - Lawrenceville, New Jersey
  - New Brunswick, New Jersey
  - Princeton, New Jersey
  - Albuquerque, New Mexico
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wexford, Pennsylvania
  - Columbia, South Carolina
  - Sioux Falls, South Dakota
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Burlington, Vermont
  - Norfolk, Virginia
  - Richmond, Virginia
  - Renton, Washington
  - Seattle, Washington

REFERENCES:
- [Result] Sutter G, Schmelter T, Gude K, Schaefers M, Gerlinger C, Archer DF. Population pharmacokinetic/pharmacodynamic evaluation of low-dose drospirenone with 17beta-estradiol in postmenopausal women with moderate to severe vasomotor symptoms. Menopause. 2014 Mar;21(3):236-42. doi: 10.1097/GME.0b013e31829c12e8. PMID 23963309
- [Result] Archer DF, Schmelter T, Schaefers M, Gerlinger C, Gude K. A randomized, double-blind, placebo-controlled study of the lowest effective dose of drospirenone with 17beta-estradiol for moderate to severe vasomotor symptoms in postmenopausal women. Menopause. 2014 Mar;21(3):227-35. doi: 10.1097/GME.0b013e31829c1431. PMID 23963307
- [Result] K. Gude; T. Schmelter; M. Schaefers; C. Gerlinger. Efficacy of low dose Angeliq (0.5 mg E2 and 0.25 or 0.5 mg DRSP) compared to Angeliq (1 mg E2 and 1, 2 or 3 mg DRSP) in postmenopausal women with moderate to severe hot flushes. Menopause, Vol. 19, No. 12, 2012 * 2012, P-36, p 1388
- [Derived] Gerlinger C, Gude K, Hiemeyer F, Schmelter T, Schafers M. An empirically validated responder definition for the reduction of moderate to severe hot flushes in postmenopausal women. Menopause. 2012 Jul;19(7):799-803. doi: 10.1097/gme.0b013e31823de8ba. PMID 22228322

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 79 centers in the United States from 26 Mar 2007 (date of first participant's first visit) to 03 Nov 2008 (date of last participant's last visit)
Pre-assignment Details: 2457 Screened; 1722 Screen Failures; 735 randomized; 726 treated (Safety Analysis Set, SAF); 710 Full Analysis Set (FAS, randomized subjects with Baseline vasomotor symptom (VMS) data, took ≥1 study dose plus ≥1 VMS data day postdose); 569 Per Protocol Set (PPS, all subjects in FAS with ≥75% study drug compliance and no major protocol violations).
Period: Overall Study
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Started | 183 | 184 | 185 | 183
Participants Received Treatment | 181 (SAF=all randomized participants who took at least 1 dose of study medication.) | 183 (SAF=all randomized participants who took at least 1 dose of study medication.) | 182 (SAF=all randomized participants who took at least 1 dose of study medication.) | 180 (SAF=all randomized participants who took at least 1 dose of study medication.)
Baseline and Postdose VMS Data Available | 178 (FAS=all randomized participants with Baseline VMS data and at least 1 day VMS data postdose.) | 177 (FAS=all randomized participants with Baseline VMS data and at least 1 day VMS data postdose.) | 179 (FAS=all randomized participants with Baseline VMS data and at least 1 day VMS data postdose.) | 176 (FAS=all randomized participants with Baseline VMS data and at least 1 day VMS data postdose.)
Completed | 160 | 164 | 158 | 153
Not Completed | 23 | 20 | 27 | 30
Not completed — Adverse Event | 7 | 4 | 6 | 4
Not completed — Lost to Follow-up | 4 | 5 | 2 | 6
Not completed — Protocol Violation | 1 | 2 | 1 | 3
Not completed — Withdrawal by Subject | 2 | 5 | 9 | 10
Not completed — Site termination | 2 | 0 | 0 | 1
Not completed — Randomization in Error | 2 | 0 | 1 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 1
Not completed — Non-compliant with study drug | 1 | 0 | 5 | 0
Not completed — Non-compliant with visit schedule | 1 | 1 | 1 | 2
Not completed — Hormone fear | 0 | 0 | 0 | 1
Not completed — Lost interest in study participation | 0 | 1 | 0 | 0
Not completed — In-/Exclusion criterion violated | 2 | 1 | 2 | 1
Not completed — Move | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo | Total
Number analyzed (Participants) | 178 | 177 | 179 | 176 | 710
Age, Continuous [Mean (Standard Deviation); unit: years] — The population included all randomized participants with Baseline VMS data and at least 1 day VMS data postdose. Full Analysis Set (FAS).
  years | 53.8 (5.61) | 53.5 (5.77) | 53.3 (6.05) | 53.4 (6.46) | 53.5 (5.97)
Sex: Female, Male [Count of Participants; unit: Participants] — The population included all randomized participants with Baseline VMS data and at least 1 day VMS data postdose. Full Analysis Set (FAS).
  Participants
    Female | 178 | 177 | 179 | 176 | 710
    Male | 0 | 0 | 0 | 0 | 0
Number of participants with hysterectomy/oophorectomy [Number; unit: Participants] — The population included all randomized participants with Baseline VMS data and at least 1 day VMS data postdose. Full Analysis Set (FAS).
  Participants
    hysterectomized | 98 | 91 | 98 | 99 | 386
    oophorectomized | 61 | 61 | 63 | 59 | 244
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/sqm] — The population included all randomized participants with Baseline VMS data and at least 1 day VMS data postdose. Full Analysis Set (FAS).
  kg/sqm | 29.070 (6.0636) | 28.190 (5.6965) | 29.080 (5.7410) | 27.882 (5.7859) | 28.543 (5.8370)
Years since last menstruation at baseline [Mean (Standard Deviation); unit: years] — The population included all randomized participants with Baseline VMS data and at least 1 day VMS data postdose. Full Analysis Set (FAS).
  years | 9.913 (8.6719) | 8.784 (7.9947) | 9.214 (8.1892) | 9.509 (8.9693) | 9.355 (8.4560)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Weekly Frequency of Moderate to Severe Hot Flushes (Median Value)
Description: Subjects record daily on the diary cards the frequency and severity of hot flushes during the treatment period as none, mild, moderate or severe. Absolute change calculated as week 12 number of moderate to severe hot flushes minus baseline number.
Time Frame: Baseline until 12 weeks of treatment
Population: Full analysis set (Intention to Treat (ITT)) with last observation carried forward approach (LOCF). Numbers differ from the complete full analysis set due to missing Week 1 data.
Measure: Median (Full Range); unit: Hot Flushes per week
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 177 | 175 | 178 | 176
Hot Flushes per week | -54.515 [-324.6 to 60.82] | -54.125 [-215.9 to 9.03] | -44.389 [-145.4 to 91.25] | -30.020 [-485.3 to 55.91]
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.5mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 12 in the number of hot flushes is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/van Elteren — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; stratification by center
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.25mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 12 in the number of hot flushes is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/van Elteren — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; stratification by center
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison between E2 (0.3mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 12 in the number of hot flushes is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p = 0.0005, Wilcoxon/van Elteren — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; stratification by center

2. Primary Outcome: Change From Baseline to Week 4 in Weekly Frequency of Moderate to Severe Hot Flushes (Median Value)
Description: Subjects record daily on the diary cards the frequency and severity of hot flushes during the treatment period as none, mild, moderate or severe. Absolute change calculated as week 4 number of moderate to severe hot flushes minus baseline number.
Time Frame: Baseline until 4 weeks of treatment
Population: Full analysis set (ITT) with last observation carried forward approach (LOCF). Numbers differ from the complete full analysis set due to missing Week 1 data.
Measure: Median (Full Range); unit: Hot Flushes per week
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 177 | 174 | 177 | 176
Hot Flushes per week | -46.868 [-276.63 to 60.82] | -37.596 [-162.15 to 35.00] | -31.621 [-141.44 to 37.91] | -15.109 [-666.33 to 27.17]
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.5mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 4 in the number of hot flushes is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/ van Elteren — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; stratification by center
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.25mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 4 in the number of hot flushes is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/van Elteren — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; stratification by center
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison between E2 (0.3mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 4 in the number of hot flushes is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/van Elteren — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; stratification by center

3. Primary Outcome: Change From Baseline to Week 12 in Weekly Mean Daily Severity of Moderate to Severe Hot Flushes (Median Value)
Description: Subjects record daily on the diary cards the frequency and severity of hot flushes during the treatment period as none, mild, moderate or severe. Daily score is calculated as [(2 x number of moderate hot flushes) + (3 x number of severe hot flushes)] / (total number of moderate to severe hot flushes on that day). Range = 0 (lowest severity) to 3 (highest severity). Absolute change calculated as week 12 severity of moderate to severe hot flushes minus baseline severity.
Time Frame: Baseline until 12 weeks of treatment
Population: as for outcome 2
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 177 | 175 | 178 | 176
Scores on a scale | -1.9294 [-3.000 to 0.480] | -1.000 [-3.000 to 0.443] | -0.2638 [-3.000 to 0.337] | -0.0698 [-3.000 to 0.542]
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.5mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 12 in the mean daily severity of hot flushes is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/van Elteren — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; stratification by center
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.25mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 12 in the mean daily severity of hot flushes is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/van Elteren — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; stratification by center
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison between E2 (0.3mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 12 in the mean daily severity of hot flushes is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p = 0.0096, Wilcoxon/van Elteren — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; stratification by center

4. Primary Outcome: Change From Baseline to Week 4 in Weekly Mean Daily Severity of Moderate to Severe Hot Flushes (Median Value)
Description: Subjects record daily on the diary cards the frequency and severity of hot flushes during the treatment period as none, mild, moderate or severe. Daily score is calculated as [(2 x number of moderate hot flushes) + (3 x number of severe hot flushes)] / (total number of moderate to severe hot flushes on that day). Range = 0 (lowest severity) to 3 (highest severity). Absolute change calculated as week 4 severity of moderate to severe hot flushes minus baseline severity.
Time Frame: Baseline until 4 weeks of treatment
Population: as for outcome 2
Measure: Median (Full Range); unit: Scorese on a scale
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 177 | 174 | 177 | 176
Scorese on a scale | -0.2905 [-3.000 to 0.383] | -0.1821 [-2.800 to 1.267] | -0.0651 [-2.898 to 0.380] | 0.0000 [-3.000 to 0.516]
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.5mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 4 in the mean daily severity of hot flushes is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/van Elteren — Significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; Stratification by center
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.25mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 4 in the mean daily severity of hot flushes is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/van Elteren — Significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; Stratification by center
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison between E2 (0.3mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 4 in the mean daily severity of hot flushes is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p = 0.0005, Wilcoxon/van Elteren — Significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; Stratification by center

5. Secondary Outcome: Change From Baseline to Week 12 in Vaginal pH
Description: Vaginal pH determined following speculum examination using vaginal pH paper and recorded on case report form (CRF). Absolute change calculated as week 12 pH minus baseline pH.
Time Frame: Baseline until 12 weeks of treatment
Population: Full analysis set (ITT). Numbers differ from the complete full analysis set due to missing data.
Measure: Mean (Standard Deviation); unit: (pH)
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 167 | 169 | 169 | 158
(pH) | -0.63 (0.874) | -0.63 (0.935) | -0.66 (0.967) | -0.06 (0.698)
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.5mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 12 in vaginal pH is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/van Elteren; Stratification by center
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.25mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 12 in vaginal pH is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/van Elteren; Stratification by center
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison between E2 (0.3 mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 12 in vaginal pH is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/van Elteren; Stratification by center

6. Secondary Outcome: Change From Baseline to Week 12 in Vaginal Maturation Value
Description: Calculated as (percentage of superficial cells) + 0.5 * (percentage of intermediate cells). Absolute change calculated as week 12 value minus baseline value.
Time Frame: Baseline until 12 weeks of treatment
Population: Full analysis set (ITT). Numbers differ from the complete full analysis set due to missing data.
Measure: Mean (Standard Deviation); unit: Percentages of cells
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 161 | 170 | 164 | 157
Percentages of cells | 10.07 (28.638) | 11.71 (29.185) | 7.69 (25.627) | -2.41 (20.923)
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.5mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 12 in vaginal maturation value is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/van Elteren; stratification by center
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.25mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 12 in vaginal maturation value is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/van Elteren; Stratification by center
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison between E2 (0.3mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The distribution of the change from baseline to week 12 in vaginal maturation value is identical in both arms, alternative: there is a shift in the distribution; Test type: Superiority or Other; p < 0.0001, Wilcoxon/van Elteren; Stratification by center

7. Secondary Outcome: Symptoms of Vulvar and Vaginal Atrophy: Severity of Symptom 'Vaginal Dryness'
Description: Subjects self-assessed symptom severity
Time Frame: After 12 weeks of treatment
Population: Full analysis set. Numbers differ from the complete full analysis set due to missing data.
Measure: Number; unit: participants
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 172 | 171 | 172 | 164
participants
  none | 83 | 70 | 71 | 70
  mild | 59 | 52 | 62 | 47
  moderate | 24 | 38 | 29 | 35
  severe | 6 | 11 | 10 | 12
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.0314, Cochran-Mantel-Haenszel — no correction for multiplicity; stratification by center
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.8780, Cochran-Mantel-Haenszel; Stratification by center
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.5908, Cochran-Mantel-Haenszel; Stratification by center

8. Secondary Outcome: Symptoms of Vulvar and Vaginal Atrophy: Severity of Symptom 'Vaginal and/or Vulvar Irritation/Itching'
Description: Subjects self-assessed symptom severity
Time Frame: After 12 weeks of treatment
Population: Full analysis set. Numbers differ from the complete full analysis set due to missing data.
Measure: Number; unit: participants
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 172 | 171 | 172 | 164
participants
  none | 152 | 140 | 146 | 128
  mild | 20 | 24 | 21 | 22
  moderate | 0 | 3 | 5 | 11
  severe | 0 | 4 | 0 | 3
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.0027, Cochran-Mantel-Haenszel — no correction for multiplicity; Stratification by center
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.4463, Cochran-Mantel-Haenszel; Stratification by center
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.0303, Cochran-Mantel-Haenszel; Stratification by center

9. Secondary Outcome: Symptoms of Vulvar and Vaginal Atrophy: Severity of Symptom 'Dysuria'
Description: Subjects self-assessed symptom severity
Time Frame: After 12 weeks of treatment
Population: Full analysis set. Numbers differ from the complete full analysis set due to missing data.
Measure: Number; unit: participants
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 172 | 171 | 170 | 162
participants
  none | 166 | 169 | 167 | 153
  mild | 6 | 2 | 1 | 9
  moderate | 0 | 0 | 1 | 0
  severe | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.4397, Cochran-Mantel-Haenszel — no correction for multiplicity; Stratification by center
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.0132, Cochran-Mantel-Haenszel; Stratification by center
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.3250, Cochran-Mantel-Haenszel; Stratification by center

10. Secondary Outcome: Symptoms of Vulvar and Vaginal Atrophy: Severity of Symptom 'Vaginal Pain Associated With Sexual Activity'
Description: Subjects self-assessed symptom severity
Time Frame: After 12 weeks of treatment
Population: Full analysis set. Numbers differ from the complete full analysis set due to missing data.
Measure: Number; unit: participants
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 166 | 165 | 162 | 152
participants
  none | 128 | 132 | 127 | 118
  mild | 21 | 22 | 21 | 19
  moderate | 13 | 7 | 11 | 11
  severe | 4 | 4 | 3 | 4
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.9555, Cochran-Mantel-Haenszel — no correction for multiplicity; Stratification by center
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.1743, Cochran-Mantel-Haenszel; Stratification by center
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.4395, Cochran-Mantel-Haenszel; Stratification by center

11. Secondary Outcome: Symptoms of Vulvar and Vaginal Atrophy: Severity of Symptom 'Vaginal Bleeding Associated With Sexual Activity'
Description: Subjects self-assessed symptom severity
Time Frame: After 12 weeks of treatment
Population: Full analysis set. Numbers differ from the complete full analysis set due to missing data.
Measure: Number; unit: participants
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 166 | 165 | 162 | 153
participants
  none | 164 | 162 | 159 | 151
  mild | 2 | 2 | 3 | 2
  moderate | 0 | 1 | 0 | 0
  severe | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.8966, Cochran-Mantel-Haenszel — no correction for multiplicity; Stratification by center
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.7512, Cochran-Mantel-Haenszel; Stratification by center
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison of active treatment arm with placebo on complete 2*4 table; Test type: Superiority or Other; p = 0.8751, Cochran-Mantel-Haenszel; Stratification by center

12. Secondary Outcome: Urogenital Symptoms: Number of Participants With Symptom 'Frequent Urination'
Description: Subjects self-assessed presence or absence of symptom
Time Frame: After 12 weeks of treatment
Population: Full analysis set (ITT). Numbers differ from the complete full analysis set due to missing data.
Measure: Number; unit: participants
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 173 | 171 | 172 | 163
participants | 45 | 56 | 62 | 57
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo; Test type: Superiority or Other; p = 0.1067, Cochran-Mantel-Haenszel; Stratification for center
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo; Test type: Superiority or Other; p = 0.6011, Cochran-Mantel-Haenszel; Stratification for center
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison of active treatment arm with placebo; Test type: Superiority or Other; p = 0.4408, Cochran-Mantel-Haenszel; Stratification for center

13. Secondary Outcome: Urogenital Symptoms: Number of Participants With Symptom 'Involuntary Urination When Laughing or Coughing'
Description: Subjects self-assessed presence or absence of symptom
Time Frame: After 12 weeks of treatment
Population: Full analysis set (ITT). Numbers differ from the complete full analysis set due to missing data.
Measure: Number; unit: participants
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 172 | 170 | 172 | 164
participants | 70 | 53 | 53 | 48
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo; Test type: Superiority or Other; p = 0.0144, Cochran-Mantel-Haenszel; Stratification for center
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo; Test type: Superiority or Other; p = 0.5589, Cochran-Mantel-Haenszel; Stratification for center
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison of active treatment arm with placebo; Test type: Superiority or Other; p = 0.5500, Cochran-Mantel-Haenszel; Stratification for center

14. Secondary Outcome: Urogenital Symptoms: Number of Participants With Symptom 'Urination at Night'
Description: Subjects self-assessed presence or absence of symptom; and if present recorded average number of times per night: 1; 2 to 4; more than 4.
Time Frame: After 12 weeks of treatment
Population: Full analysis set (ITT). Numbers differ from the complete full analysis set due to missing data.
Measure: Number; unit: participants
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 173 | 171 | 172 | 164
participants | 99 | 114 | 114 | 111
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo; Test type: Superiority or Other; p = 0.2179, Cochran-Mantel-Haenszel; Stratification for center
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison of active treatment arm with placebo; Test type: Superiority or Other; p = 0.7749, Cochran-Mantel-Haenszel; Stratification for center
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison of active treatment arm with placebo; Test type: Superiority or Other; p = 0.8307, Cochran-Mantel-Haenszel; Stratification for center

15. Other Pre Specified Outcome: Change From Baseline to Week 12 in Weekly Frequency of Moderate to Severe Hot Flushes (Mean Value)
Description: as for outcome 1
Time Frame: Baseline until 12 weeks of treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hot Flushes per week
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 177 | 175 | 178 | 176
Hot Flushes per week | -60.331 (37.5217) | -55.317 (30.2311) | -41.783 (32.6122) | -31.916 (44.4507)
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.5mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The mean change from baseline to week 12 is identical in both arms, alternative: there is a difference in the mean change from baseline; Test type: Superiority or Other; p < 0.0001, ANCOVA — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; treatment, center and baseline value used as covariate; Mean Difference (Final Values) = -27.6, 95% CI [-33.2 to -22.0] — Change in active treatment arm minus change in placebo arm
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.25mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The mean change from baseline to week 12 is identical in both arms, alternative: there is a difference in the mean change from baseline; Test type: Superiority or Other; p < 0.0001, ANCOVA — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; treatment, center and baseline value used as covariate; Mean Difference (Final Values) = -22.2, 95% CI [-27.8 to -16.6] — Change in active treatment arm minus change in placebo arm
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison between E2 (0.3mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The mean change from baseline to week 12 is identical in both arms, alternative: there is a difference in the mean change from baseline; Test type: Superiority or Other; p = 0.0007, ANCOVA — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; treatment, center and baseline value used as covariate; Mean Difference (Final Values) = -9.8, 95% CI [-15.4 to -4.2] — Change in active treatment arm minus change in placebo arm

16. Other Pre Specified Outcome: Change From Baseline to Week 4 in Weekly Frequency of Moderate to Severe Hot Flushes (Mean Value)
Description: as for outcome 2
Time Frame: Baseline until 4 weeks of treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hot Flushes per week
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 177 | 174 | 177 | 176
Hot Flushes per week | -48.810 (35.7876) | -38.989 (27.7812) | -32.633 (28.1349) | -24.195 (54.7480)
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.5mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The mean change from baseline to week 4 is identical in both arms, alternative: there is a difference in the mean change from baseline; Test type: Superiority or Other; p < 0.0001, ANCOVA — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; treatment, center and baseline value used as covariate; Mean Difference (Final Values) = -23.9, 95% CI [-29.9 to 17.8] — Change in active treatment arm minus change in placebo arm
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; Comparison between DRSP/E2 (0.25mg/0.5mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The mean change from baseline to week 4 is identical in both arms, alternative: there is a difference in the mean change from baseline; Test type: Superiority or Other; p < 0.0001, ANCOVA — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; treatment, center and baseline value used as covariate; Mean Difference (Final Values) = -14.2, 95% CI [-20.2 to -8.1] — Change in active treatment arm minus change in placebo arm
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison between E2 (0.3mg) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The mean change from baseline to week 4 is identical in both arms, alternative: there is a difference in the mean change from baseline; Test type: Superiority or Other; p = 0.0054, ANCOVA — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; treatment, center and baseline value used as covariate; Mean Difference (Final Values) = -8.6, 95% CI [-14.6 to -2.5] — Change in active treatment arm minus change in placebo arm

17. Other Pre Specified Outcome: Change From Baseline to Week 12 in Weekly Mean Daily Severity of Moderate to Severe Hot Flushes (Mean Value)
Description: Subjects record daily on the diary cards the frequency and severity of hot flushes during the treatment period as none, mild, moderate or severe. Daily score is calculated as [(2 x number of moderate hot flushes) + (3 x number of severe hot flushes)] / (total number of moderate to severe hot flushes on that day). Range = 0 (lowest severity) to 3 (highest severity). Absolute change calculated as week 12 severity moderate to severe hot flushes minus baseline severity.
Time Frame: Baseline until 12 weeks of treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 177 | 175 | 178 | 176
Scores on a scale | -1.4473 (1.11616) | -1.2141 (1.08299) | -0.7822 (1.03497) | -0.3873 (0.76950)
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; treatment, center and baseline value used as covariate; Mean Difference (Final Values) = -1.069, 95% CI [-1.280 to -0.859] — Change in active treatment arm minus change in placebo arm
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; treatment, center and baseline value used as covariate; Mean Difference (Final Values) = -0.803, 95% CI [-1.013 to -0.593] — Change in active treatment arm minus change in placebo arm
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; [analysis description as in outcome 15, analysis 3]; Test type: Superiority or Other; p = 0.0007, ANCOVA — significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; treatment, center and baseline value used as covariate; Mean Difference (Final Values) = -0.361, 95% CI [-0.570 to -0.152] — Change in active treatment arm minus change in placebo arm

18. Other Pre Specified Outcome: Change From Baseline to Week 4 in Weekly Mean Daily Severity of Moderate to Severe Hot Flushes (Mean Value)
Description: Subjects record daily on the diary cards the frequency and severity of hot flushes during the treatment period as none, mild, moderate or severe. Daily score is calculated as [(2 x number of moderate hot flushes) + (3 x number of severe hot flushes)] / (total number of moderate to severe hot flushes on that day). Range = 0 (lowest severity) to 3 (highest severity). Absolute change calculated as week 4 severity moderate to severe hot flushes minus baseline severity.
Time Frame: Baseline until 4 weeks of treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Number analyzed (Participants) | 177 | 174 | 177 | 176
scores on a scale | -0.8347 (1.02226) | -0.5859 (0.89106) | -0.4033 (0.73774) | -0.1926 (0.63585)
Statistical Analysis 1: Comparison: 0.5mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; Treatment, Center, and Baseline value used as covariate; Mean Difference (Final Values) = -0.635, 95% CI [-0.813 to -0.458]
Statistical Analysis 2: Comparison: 0.25mg DRSP / 0.5mg E2 (BAY86-4891) vs Placebo; [analysis description as in outcome 16, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; Treatment, Center, and Baseline value used as covariate; Mean Difference (Final Values) = -0.382, 95% CI [-0.560 to -0.205]
Statistical Analysis 3: Comparison: Estradiol (E2 0.3mg) vs Placebo; Comparison between E2 (0.3) and Placebo with respect to a shift in the distribution of the end point. Null hypothesis: The mean change from baseline to week 4 is identical in both arms, alternative: there is a difference in the mean change from baseline; Test type: Superiority or Other; p = 0.0233, ANCOVA — Significance level of 1.7% is used to adjust (Bonferroni) for the comparison of three active arms with Placebo; Treatment, Center, and Baseline value used as covariate; Mean Difference (Final Values) = -0.204, 95% CI [-0.381 to -0.028]

ADVERSE EVENTS:
Arm/Group | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) | Estradiol (E2 0.3mg) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/181 | 1/183 | 3/182 | 1/180
Other Adverse Events (participants affected / at risk) | 80/181 | 75/183 | 68/182 | 64/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) (N=181) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) (N=183) | Estradiol (E2 0.3mg) (N=182) | Placebo (N=180)
Salpingitis (Infections and infestations) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.5mg DRSP / 0.5mg E2 (BAY86-4891) (N=181) | 0.25mg DRSP / 0.5mg E2 (BAY86-4891) (N=183) | Estradiol (E2 0.3mg) (N=182) | Placebo (N=180)
Nausea (Gastrointestinal disorders) | 5 | 6 | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 8 | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 4 | 0 | 3 | 1
Vomiting (Gastrointestinal disorders) | 5 | 0 | 0 | 0
Oedema peripheral (General disorders) | 2 | 4 | 0 | 1
Vaginitis bacterial (Infections and infestations) | 7 | 3 | 7 | 7
Nasopharyngitis (Infections and infestations) | 4 | 6 | 4 | 6
Urinary tract infection (Infections and infestations) | 5 | 4 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 6 | 3 | 4 | 3
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 5 | 4 | 1
Vulvovaginal candidiasis (Infections and infestations) | 2 | 5 | 1 | 0
Low density lipoprotein increased (Investigations) | 4 | 7 | 7 | 9
C-reactive protein increased (Investigations) | 2 | 6 | 3 | 4
Blood glucose increased (Investigations) | 4 | 2 | 3 | 4
Blood cholesterol increased (Investigations) | 2 | 3 | 4 | 2
Blood triglycerides increased (Investigations) | 4 | 2 | 1 | 3
Weight decreased (Investigations) | 4 | 2 | 2 | 2
Weight increased (Investigations) | 2 | 4 | 1 | 3
Gamma-glutamyltransferase increased (Investigations) | 3 | 2 | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 2 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5 | 3 | 1
Headache (Nervous system disorders) | 8 | 11 | 10 | 9
Mood swings (Psychiatric disorders) | 4 | 2 | 2 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 2 | 8 | 5 | 7
Breast tenderness (Reproductive system and breast disorders) | 12 | 6 | 1 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 4 | 3 | 5 | 5
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 4 | 2 | 1 | 1
Breast pain (Reproductive system and breast disorders) | 4 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 1 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
(A) PI will provide copy to Sponsor at least (30) days prior to date of planned submission or presentation. Sponsor will have thirty (30) days to review and provide feedback. If proposed publication presents material adverse effect on the confidentiality of Sponsor's information, then PI shall delay or prevent such publication. (B) In a multi-center trial, the investigative data will be pooled and published as a collaborative effort with consent from all parties including the Sponsor.